CLINICAL TRIAL: NCT07192614
Title: A Phase I/II Open-label, Dose Escalation and Dose Expansion Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Efficacy of AZD6621, a T Cell-engaging Antibody That Targets STEAP2, CD3, and CD8 in Adult Participants With Metastatic Prostate Cancer
Brief Title: A Study to Learn How Safe AZD6621 is, How Well it Works, and How it Moves Throughout the Body Over Time, in Adult Male Participants With Metastatic Prostate Cancer
Acronym: ACTIVATED-4-PC
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D8020C00003; 2025-520626-37 (EudraCT Number)
Record Dates: First submitted 2025-07-11; First posted 2025-09-25 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Metastatic Prostate Cancer; Prostate Cancer; Prostate Adenocarcinoma; T Cell-engaging Antibody; STEAP2; CD3; CD8
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a first in human, multicenter, open-label, dose-escalation and dose-expansion study. The study includes 2 Modules; Module 1 is investigating AZD6621 given on its own by one method of administration, and Module 2 is investigating AZD6621 on its own by a different method of administration. The study also has 2 parts: Part A Dose Escalation and Part B Dose Expansion. Part B Dose expansion will assess at least 2 doses or dosing schedules in either module. Participants will be randomised in Part B to one of these cohorts whenever possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Module 1 - Part A (Dose Escalation) (Experimental): AZD6621 Monotherapy - Administration route 1
  Interventions: Drug: AZD6621
- Module 2 - Part A (Dose Escalation) (Experimental): AZD6621 Monotherapy - Administration route 2
  Interventions: Drug: AZD6621
- Module 1/2 - Part B1 (Dose Expansion) (Experimental): AZD6621 Monotherapy - Administration route 1 (Module 1) or administration route 2 (Module 2) at Recommended Dose for Expansion 1 (RDE1)
  Interventions: Drug: AZD6621
- Module 1/2 - Part B2 (Dose Expansion) (Experimental): AZD6621 Monotherapy - Administration route 1 (Module 1) or administration route 2 (Module 2) at Recommended Dose for Expansion 2 (RDE2)
  Interventions: Drug: AZD6621

INTERVENTIONS:
Drug: AZD6621 — A T Cell-engaging Antibody that targets STEAP2, CD3, and CD8

SUMMARY:
This study is being conducted to learn more about the safety, tolerability, and effectiveness of an experimental treatment for metastatic prostate cancer called AZD6621. The study is split into different modules which will look at AZD6621 delivered by different methods. The study is also further split into 2 parts, Part A which will test different dose levels of AZD6621 to determine which doses are the best in terms of safety and side effects (dose escalation), and Part B will further test at least two AZD6621 doses in a larger group of participants (dose expansion).

DETAILED DESCRIPTION:
This is a first in human, modular, Phase I/II, open-label, multicenter study of AZD6621, in adult participants with metastatic prostate cancer. The study will consist of study modules, each evaluating safety, tolerability, PK, pharmacodynamics, and anti-tumor activity of AZD6621 in metastatic prostate cancer. The study will also characterize the PK and immunogenicity of AZD6621.

ELIGIBILITY:
Inclusion Criteria

1. Capable of giving signed informed consent and complying to the study protocol.
2. Provision of signed and dated written Optional Genomics Initiative Research Information and Consent Form.
3. ≥ 18 years of age at the time of signing the informed consent form.
4. Participants with:

   1. Histologically confirmed diagnosis of metastatic adenocarcinoma of the prostate
   2. Surgically or medically castrated, with serum testosterone levels ≤ 50 ng/dL (≤ 1.75 nmol/L) ≤ 28 days before first dose of study intervention. Participants without prior surgical castration must be currently taking and willing to continue LHRH agonist or antagonist therapy throughout the duration of the study intervention.
   3. Castration-resistant prostate cancer as defined by disease progression despite castration by orchiectomy or ongoing ADT.
   4. PSA at screening visit ≥ 1 ng/mL.
5. Provision of baseline fresh or archival tumor biopsy of prostate carcinoma is mandatory.
6. Evidence of disease progression within 6 months prior to screening with at least one of the following:

   1. PSA progression defined by a minimum of 3 rising PSA levels with an interval of ≥ 1 week between each determination.
   2. Radiographic progression of soft tissue disease by RECIST v1.1 criteria with or without PSA progression.
   3. Radiographic progression of bone metastasis by PCWG3 criteria with 2 or more documented new bone lesions on a bone scan with or without PSA progression.
7. Part A: Module 1 and Module 2:

   1. Part A: Module 1 and Module 2 prior anti-cancer treatment requirements as stated in study protocol
   2. Pharmacodynamic backfill cohort(s) only: lesion amenable for biopsy and be willing to undergo biopsy, distinct from any target lesion used in the RECIST v1.1 evaluation, unless there are no other lesions available for biopsy.
8. Part B: Module 1 and Module 2:

   1. Part B: Module 1 and Module 2 prior anti-cancer treatment requirements as stated in study protocol.
   2. Participants may have received PARP inhibitors or checkpoint inhibitors per local treatment guidelines.
   3. Sampling Requirements as stated in study protocol.
9. ECOG PS score of 0 or 1.
10. Minimum life expectancy of > 12 weeks.
11. Adequate hematological, renal, bone marrow, and liver function as documented in the protocol.
12. Body weight ≥ 35 kg.
13. Male, as assigned at birth, inclusive of all gender identities.
14. Contraceptive use by participants or participant partners as documented in the protocol and consistent with local regulations.

Exclusion Criteria

1. Any evidence of diseases (such as severe or uncontrolled systemic diseases) which in the Investigator's opinion makes it undesirable for the participant to participate in the study.
2. One or more of the following:

   1. Mean resting corrected QT interval > 470 ms,
   2. History of QT prolongation associated with other medications that required discontinuation of that medication, or any current concomitant medication known to prolong the QT interval and cause Torsades de Pointes.
   3. Congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives.
   4. Inadequate cardiac function of LVEF < 50% on screening cardiac MUGA or ECHO.
3. Cardiac arrhythmias (such as multifocal premature ventricular contractions, bigeminy, trigeminy, ventricular tachycardia), which are symptomatic or require treatment unless controlled by pacemaker; symptomatic or uncontrolled atrial fibrillation despite treatment, or asymptomatic sustained ventricular tachycardia.
4. History of another primary malignancy except for malignancy treated with curative intent with no known active disease (≥ 2 years) before the first dose of study intervention and of low potential risk for recurrence.
5. History of, or planned organ or allogeneic stem cell transplantation.
6. Unresolved toxicity from prior anti-cancer therapy of CTCAE Grade ≥ 2 (exceptions listed in protocol).
7. History of Grade ≥ 3 CRS or Grade ≥ 2 ICANS based on ASTCT criteria with prior therapy. CRS must be resolved prior to screening.
8. Previous history of hemophagocytic lymphohistiocytosis/ macrophage activation syndrome.
9. Active or prior documented autoimmune or inflammatory disorders (examples in protocol) within the past 3 years prior to the start of treatment or requiring permanent immunosuppressive therapy.
10. Spinal cord compression unless asymptomatic and treated and stable and not requiring continuous corticosteroids at a dose of > 10 mg prednisone/day or equivalent.
11. CNS pathology (examples in protocol).
12. Active or uncontrolled hepatitis B or C virus infection (exceptions listed in the protocol).
13. Known HIV infection that is not well controlled (definition for HIV infection that is well controlled is listed in protocol).
14. Radiation therapy within 4 weeks of first dose of study intervention (or local or focal radiotherapy within 2 weeks of first dose).
15. Prior anti-cancer drug exposure requirement as stated in study protocol
16. Previous anti-cancer treatment requirements as stated in study protocol
17. Systemic corticosteroids at doses exceeding 10 mg/day of prednisone or equivalent < 7 days prior to first dose.
18. Major surgical procedure or significant traumatic injury within 4 weeks prior to first dose.
19. Receipt of the last dose of anti-cancer therapy or participation in another clinical study with last dose administered in the last 21 days or 5 half-lives, whichever is shorter

    - CAR-T cell therapy within the last 6 months prior to enrolment on this study.
20. Participants with a known hypersensitivity to AZD6621 or any of its excipients.
21. Involvement in the planning and/or conduct of the study.
22. Participant is unlikely to comply with study procedures, restrictions, and requirements (as judged by the Investigator).
23. Receipt of live attenuated vaccine within 30 days prior to the first dose of study intervention or receipt of COVID-19 vaccination within 72 hours prior to the first dose of study intervention.
24. Previous enrolment in the present study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male, as assigned at birth, inclusive of all gender identities
Enrollment: 52 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2029-03-29 (Estimated); Study Completion 2029-03-29 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AE), adverse events of special interest (AESI), and serious adverse events (SAE) | From time of Informed Consent to 90 days post last dose of study intervention (up to 3 years)
  • Number of participants with AEs, AESIs, SAEs, including AEs leading to discontinuation of study intervention and clinically significant alterations from baseline in laboratory parameters, vital signs, ECGs and physical examination results
Number of participants with dose-limiting toxicity (DLT), as defined in the protocol (Part A only) | From first study dose to 21 to 28 days post first dose
  • A DLT is a toxicity defined by the study protocol that occurs from the first dose of study intervention up to the end of the DLT evaluation period that is assessed as clearly unrelated to the primary disease or intercurrent illness.
Preliminary anti-tumour activity of AZD6621 (PSA Response Rate) (Part B only) | Up to 3 years
  • Number of participants with a PSA response rate

SECONDARY OUTCOMES:
Preliminary anti-tumour activity of AZD6621 (PSA Response rate) (Part A only) | Up to 3 years
  • Number of participants with a PSA response rate
Preliminary anti-tumour activity of AZD6621 (time to PSA response) | Up to 3 years
  • Time taken to achieve a PSA response
Preliminary anti-tumour activity of AZD6621 (duration of PSA response) | Up to 3 years
  • Time PSA response lasts
Preliminary anti-tumour activity of AZD6621 (durable PSA response rate) | Up to 3 years
  • Percentage of participants who have a confirmed PSA response with a duration of at least 6 months
Preliminary anti-tumour activity of AZD6621 (time to PSA progression) | Up to 3 years
  • Time taken to achieve PSA progression
Preliminary anti-tumour activity of AZD6621 (Radiological Response - RECIST) | Up to 3 years
  • Radiological response: according to RECIST v1.1 (soft tissue) and PCWG3 (bone)
Preliminary anti-tumour activity of AZD6621 (Radiological Response - Target Lesion Percentage change) | Up to 3 years
  • Percentage change in Target Lesion size according to RECIST v1.1.
Preliminary anti-tumour activity of AZD6621 (Overall Survival 12 months) | 12 months
  • Overall Survival at 12 months
Preliminary anti-tumour activity of AZD6621 (Overall Survival) | Up to 3 years
  • Median Overall Survival
Preliminary anti-tumour activity of AZD6621 (SSRE) | Up to 3 years
  • Time to first symptomatic skeletal-related events (SSRE)
Pharmacokinetics of AZD6621 (Serum concentrations) | From first dose of study intervention to 28 days post last dose of study intervention
  • Serum concentrations of the study drug.
Pharmacokinetics of AZD6621 (Cmax) | From first dose of study intervention to 28 days post last dose of study intervention
  • Maximum observed plasma concentration of the study drug (Cmax).
Pharmacokinetics of AZD6621 (AUC) | From first dose of study intervention to 28 days post last dose of study intervention
  • Area under the plasma concentration-time curve (AUC).
Pharmacokinetics of AZD6621 (Tmax) | From first dose of study intervention to 28 days post last dose of study intervention
  • The time it takes for study drug to reach the maximum concentration (Tmax).
Pharmacokinetics of AZD6621 (t1/2) | From first dose of study intervention to 28 days post last dose of study intervention
  • Terminal elimination half life of study drug (t1/2)
Immunogenicity of AZD6621 | From first dose of study intervention to 28 days post last dose of study intervention
  • The number and percentage of participants who develop detectable anti-drug antibodies (ADA).
Tumour STEAP2 expression | Up to 3 years
  • STEAP2 expression in tumour as measured by immunohistochemistry (IHC)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (5):
  - Research Site, Tampa, Florida
  - Research Site, Boston, Massachusetts
  - Research Site, Grand Rapids, Michigan
  - Research Site, Commack, New York
  - Research Site, Providence, Rhode Island
- China (3):
  - Research Site, Beijing
  - Research Site, Guangzhou
  - Research Site, Nanjing
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Hirakata-shi
  - Research Site, Kashiwa
- Research Site, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org.
  All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/